CLINICAL TRIAL: NCT02437773
Title: Neurocircuit Mechanisms of OCD Across the Lifespan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kate D. Fitzgerald, Associate Professor, Department of Psychiatry, University of Michigan, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00091368; R01MH102242-01A1 (NIH)
Record Dates: First submitted 2015-05-02; First posted 2015-05-08 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cognitive Behavioral Therapy - Adolescents (Active Comparator): 12 Cognitive-Behavioral Therapy sessions scheduled weekly over a 12-week period.
  Interventions: Behavioral: Cognitive Behavioral Therapy - Adolescents
- Stress Management Therapy - Adolescents (Other): 12 SMT sessions scheduled weekly over a 12-week period.
  After study completion, the OCD subjects who received SMT may derive benefit for non-OCD anxiety symptoms. They will be offered a 12-week course of CBT with a study therapist to directly target OCD symptoms (i.e., a partial cross-over).
  Interventions: Behavioral: Stress Management Therapy - Adolescents; Behavioral: Optional CBT - Adolescents
- Cognitive Behavioral Therapy - Adults (Active Comparator): 12 CBT sessions scheduled weekly over a 12-week period.
  Interventions: Behavioral: Cognitive Behavioral Therapy - Adults
- Stress Management Therapy - Adults (Other): 12 SMT sessions scheduled weekly over a 12-week period.
  After study completion, the OCD subjects who received SMT may derive benefit for non-OCD anxiety symptoms. They will be offered a 12-week course of CBT with a study therapist to directly target OCD symptoms (i.e., a partial cross-over).
  Interventions: Behavioral: Stress Management Therapy - Adults; Behavioral: Optional CBT - Adults
- Healthy Control - Adolescents (Other): Healthy control adolescents matched to gender, race and socioeconomic status (SES) with adolescent patients with OCD will be enrolled. These healthy adolescents will be scanned with fMRI before and after 12 weeks, but without any intervention (i.e., no therapy).
  Interventions: Other: fMRI only - Healthy Control Adolescents
- Healthy Control - Adults (Other): Healthy control adults matched to gender, race and socioeconomic status (SES) with adult patients with OCD will be enrolled. These healthy adults will be scanned with fMRI before and after 12 weeks, but without any intervention (i.e., no therapy).
  Interventions: Other: fMRI only - Healthy Control Adults
- Optional CBT - Adolescents (Other): OCD adolescent participants who were randomized to the SMT and have completed all study procedures will be offered an additional 12 weeks of Optional Cognitive-Behavioral Therapy.
  Interventions: Behavioral: Optional CBT - Adolescents
- Optional CBT - Adults (Other): OCD adult participants who were randomized to the SMT and have completed all study procedures will be offered an additional 12 weeks of Optional Cognitive-Behavioral Therapy.
  Interventions: Behavioral: Optional CBT - Adults

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy - Adolescents — A therapy which gradually yet repeatedly exposes adolescent patients to their obsessive compulsive-relevant "error" cues during a task performance until their anxiety habituates.
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy - Adolescents
Behavioral: Stress Management Therapy - Adolescents — An active control therapy with minimal effects on OCD symptoms.
  Other Names: SMT
  Arms: Stress Management Therapy - Adolescents
Behavioral: Optional CBT - Adolescents — This is the cross-over element for those that completed the SMT treatment group and opt to have the OCD treatment.
  Other Names: CBT
  Arms: Optional CBT - Adolescents; Stress Management Therapy - Adolescents
Behavioral: Cognitive Behavioral Therapy - Adults — A therapy which gradually yet repeatedly exposes adult patients to their obsessive compulsive-relevant "error" cues during a task performance until their anxiety habituates.
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy - Adults
Behavioral: Stress Management Therapy - Adults — An active control therapy with minimal effects on OCD symptoms.
  Other Names: SMT
  Arms: Stress Management Therapy - Adults
Behavioral: Optional CBT - Adults — This is the cross-over element for those that completed the SMT treatment group and opt to have the OCD treatment.
  Other Names: CBT
  Arms: Optional CBT - Adults; Stress Management Therapy - Adults
Other: fMRI only - Healthy Control Adults — Two fMRI's only, scheduled at 12-weeks apart. This is for Healthy Control Adults and is used only as a means for observation, NOT as an intervention to be studied.
  Arms: Healthy Control - Adults
Other: fMRI only - Healthy Control Adolescents — Two fMRI's only, scheduled at 12-weeks apart. This is for Healthy Control Adolescents and is used only as a means for observation, NOT as an intervention to be studied.
  Arms: Healthy Control - Adolescents

SUMMARY:
Obsessive-compulsive disorder (OCD), characterized by intrusive thoughts (obsessions) and related behavioral rituals (compulsions), is a common psychiatric illness that often emerges in childhood and causes life-long disability in over 50% of patients. Psychological theory suggests that OCD symptoms are driven by a person's difficulty disengaging their feelings from simple tasks (e.g. washing hands, locking a door) due to excessive anxiety about performance errors. Cognitive behavioral therapy (CBT), the gold standard treatment for OCD, repeatedly exposes patients to their OCD-stressor until this anxiety is reduced. While CBT is typically more effective in teenagers than adults, patients from both age groups are usually left with residual symptoms, highlighting the need for better treatments. In this study, CBT will be studied in both teen-aged and adult patients. Two groups, both with childhood onset OCD, will be randomized to either CBT for OCD or stress management training (SMT), an active therapy but with minimal effects on OCD symptoms. The investigators will also study age-matched, healthy controls as comparison subjects.

Before and after 12 weeks of CBT, all subjects will undergo functional Magnetic Resonance Imaging (fMRI) scans to see what regions of the brain become active when a concentration task is performed and how that activation is changed after CBT. The purpose of this study is to demonstrate the brain changes associated with CBT treatment and how differences in these changes in teenage compared to adult patients may drive differences in CBT response.

DETAILED DESCRIPTION:
While the study itself is of parallel design for its data-collection and measurement purpose, it is listed as a partial-crossover design in the IRB-approved protocol because subjects randomized to the SMT group are given the option of entering 12-weeks of CBT sessions after all of their SMT data collection. To understand brain changes that occur with CBT compared to SMT in both age groups, the investigators will collect fMRI data before and after therapy. Some limited data will be collected in patients who are initially randomized to SMT but then opt to crossover to CBT. fMRI data will also be collected in healthy teens and adults before and after 12 weeks (but without intervening therapy) to allow the investigators to control for the simple effects of time that may cause brain changes that are not related to therapy.

ELIGIBILITY:
Inclusion Criteria for all OCD Subjects & Healthy Volunteers:

* Male or female
* Age 13-17 (inclusive) subjects diagnosed with OCD, age of onset before 15 years
* Age 25-45 (inclusive) subjects diagnosed with OCD, age of onset before 15 years
* Age 13-17 (inclusive) year old healthy volunteers
* Age 25-45 (inclusive) year old healthy volunteers
* OCD adolescent and adult subjects can be on medications but will have to be on a stable medication regimen for at least 4 weeks prior to enrolling.
* Able and willing to give informed consent
* Ability to tolerate small, enclosed spaces without anxiety

Exclusion Criteria for OCD Subjects:

* Anyone between the ages of 18-24 (inclusive range)
* No lifetime diagnosis of bipolar or psychosis disorders
* Age of OCD onset after 15 years old
* No substance/alcohol abuse in the past 6 months
* No lifetime history of substance/alcohol dependence
* No evidence of suicidal intentions or behaviors in the past 6 months
* No history of serious medical or neurological illness
* No history of closed head injury (e.g. loss of consciousness)
* Pregnant or trying to become pregnant

Additional Exclusion Criteria for Healthy Volunteers:

* No history of past or current mental illness
* Not taking any medication, prescription or non-prescription, with psychotropic effects
* First-degree family members with OCD or tic disorders

Ages: 13 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 206 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Brain activity as assessed by Magnetic Resonance Imaging (fMRI) scans | Baseline to 12-weeks
  fMRI BOLD signal response of posterior medial frontal cortex (pMFC), ventral medial prefrontal cortex (vmPFC) and anterior insula (aIns) during performance monitoring. This signal will be measured as BOLD contrast estimates for errors compared to correct trials based on average signal in a priori defined regions of interest for pMFC, vmPFC and aIns. The investigators are looking for increases in pMFC activation in adolescents from pre- to post-treatment. In contrast, the investigators are looking for increases in inverse connectivity (resting state and during task) between vmPFC and aIns in adults from pre- to post-treatment.

SECONDARY OUTCOMES:
OCD symptom severity measured by the Yale Brown Obsessive Compulsive Scale for adults or the Child Yale Brown Obsessive Compulsive Scale for adolescents. | Baseline to 12-weeks
  OCD symptom severity measured by the Yale Brown Obsessive Compulsive Scale for adults and the Child Yale Brown Obsessive Compulsive Scale for adolescents. This scale is administered by an independent assessor to rate OCD symptom severity on a scale of 0 to 40, with 40 being most severe. The investigators are looking for decreases in OCD severity ratings from pre- to post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Fitzgerald, MD, Principal Investigator — University of Michigan, Dept of Psychiatry
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Himle JA, Grogan-Kaylor A, Hiller MA, Mannella KA, Norman LJ, Abelson JL, Prout A, Shunnarah AA, Becker HC, Russman Block SR, Taylor SF, Fitzgerald KD. Exposure and response prevention versus stress management training for adults and adolescents with obsessive compulsive disorder: A randomized clinical trial. Behav Res Ther. 2024 Jan;172:104458. doi: 10.1016/j.brat.2023.104458. Epub 2023 Dec 12. PMID 38103359
- [Derived] Rueppel M, Mannella KA, Fitzgerald KD, Schroder HS. Post-error slowing in anxiety and obsessive-compulsive disorders. Cogn Affect Behav Neurosci. 2022 Jun;22(3):610-624. doi: 10.3758/s13415-021-00976-9. Epub 2021 Dec 29. PMID 34966981
- [Derived] Norman LJ, Mannella KA, Yang H, Angstadt M, Abelson JL, Himle JA, Fitzgerald KD, Taylor SF. Treatment-Specific Associations Between Brain Activation and Symptom Reduction in OCD Following CBT: A Randomized fMRI Trial. Am J Psychiatry. 2021 Jan 1;178(1):39-47. doi: 10.1176/appi.ajp.2020.19080886. Epub 2020 Aug 28. PMID 32854533